CLINICAL TRIAL: NCT00350896
Title: Comparative Study of the Efficacy of Thumb Orthoses in the Base of the Thumb (BTOA)
Brief Title: Safety Study of Thumb Orthoses in Osteoarthritis in the Base of the Thumb (BTOA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P020916
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2006-07-11 (Estimated); Status verified 2006-01

CONDITIONS: Osteoarthritis
Keywords: trapezotrapezoidial; scaphotrapezial; thumb; pain; orthoses; Osteoarthritis in the BTOA concerns the trapezometacarpal joint
MeSH Terms: conditions — Osteoarthritis; Pain

INTERVENTIONS:
Device: Thumb orthoses

SUMMARY:
The prevalence of digital osteoarthritis varies according to whether a radiological or clinical definition is adopted.

Interventions: Thumb orthoses to be worn at night and usual care vs usual care. Outcome measures: Pain at 1 month assessed on visual analog scale is the main outcome measure. Disability at 6 months (Cochin Hand Function Scale) and deformation at 1 year are the main secondary outcome measures.

DETAILED DESCRIPTION:
The prevalence of digital osteoarthritis varies according to whether a radiological or clinical definition is adopted. Radiologically defined osteoarthritis of the hand has been estimated to represent 38% of women and 24.5% of men over 66 years of age but higher prevalence of 60-70% has also been reported. Of patients with radiological signs, 20 to 40% become symptomatic. For patients over 55 years of age, the distal interphalangeal joints are the most prevalent site of osteoarthritis (20%) determined radiologically and clinically, followed by the base of the thumb (8%) and proximal interphalangeal joints (5%). This prevalence increases with age, and the incidence peaks in perimenopausal women. Osteoarthritis in the base of the thumb (BTOA) concerns the trapeziometacarpal joint, with a possible secondary location at the trapezotrapezoidial and scaphotrapezial joints. BTOA induces a closure of the first web, which in turn causes an alteration of the thumb-index pinch and therefore a limitation in hand function. Pain induced by the compression of the thumb column during pinching could also lead to functional disability. Effect of a simple intervention such as wearing rest thumb orthoses on pain and disability is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Pain at the base of the thumb 30 mm on VAS
* Patient aged 45 and < 75 years old
* At least 2 of the 5 items on the trapeziometacarpal joint radiograph osteophytes
* joint space narrowing
* subchondral bone sclerosis
* subchondral cysts
* At least 1 of the 2 clinical items trapeziometacarpal joint enlargement closure of the first web

Exclusion Criteria:

* Post traumatic osteoarthritis
* Cristal arthropathy
* Inflammatory arthritis
* Neurologic disorder involving upper limb
* Psychiatric disorder needing treatment adaptation in the last 3 months
* Hand or wrist trauma within the last 2 months
* Previous hand surgery
* Unable to speak or write French
* Pregnancy
* Collagen diseases (Dupuytren, Marfan, Ehlers Danlos syndromes)
* Hand or wrist infiltration within 2 months
* Skin disease interfering with the wearing of the orthoses
* Having already worn a BTOA orthoses
* Having bilateral BTOA without predominant symptomatic side

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-12; Study Completion 2005-12

PRIMARY OUTCOMES:
Pain at 1 month assessed on visual analog scale is the main outcome measure.

SECONDARY OUTCOMES:
Disability at 6 months (Cochin Hand Function Scale) and deformation at 1 year are the main secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Poiraudeau, MD, Phd, Principal Investigator — Cochin Hospital AP-HP

REFERENCES:
- [Derived] Rannou F, Dimet J, Boutron I, Baron G, Fayad F, Mace Y, Beaudreuil J, Richette P, Ravaud P, Revel M, Poiraudeau S. Splint for base-of-thumb osteoarthritis: a randomized trial. Ann Intern Med. 2009 May 19;150(10):661-9. doi: 10.7326/0003-4819-150-10-200905190-00003. PMID 19451573